CLINICAL TRIAL: NCT06098001
Title: Bioavailability Study of Phenolics in Hemp Hull Dietary Fiber
Brief Title: Bioavailability Study of Hemp Phenolics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brightseed (Industry)
Collaborators: Biofortis Mérieux NutriSciences (Other); University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BIO-2311
Record Dates: First submitted 2023-10-05; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Bioavailability; Metabolites; Excretion
MeSH Terms: interventions — Dietary Fiber

STUDY DESIGN:
Intervention Model Description: Participants receive same treatment in dose escalation design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose fiber (Active Comparator): Dose esacalation design
  Interventions: Dietary Supplement: Low dose dietary fiber
- High dose of fiber (Active Comparator): Dose escalation design which is one arm with low and followed by high dose
  Interventions: Dietary Supplement: High dose dietary fiber

INTERVENTIONS:
Dietary Supplement: Low dose dietary fiber — Subjects will receive a low dose or high dose of the dietary fiber product in a dose esacalation design
  Arms: Low dose fiber
Dietary Supplement: High dose dietary fiber — Subjects will receive a low dose or high dose of the dietary fiber product in a dose escalation design
  Arms: High dose of fiber

SUMMARY:
The aim is to determine the bioavailability of the polyphenol fraction form a commercially available hemp hull fiber at two different amounts in generally healthy adults. Additional objectives include determining specific metabolites produced over a 24 to 48-hour period following the hemp fiber consumption. Subjects will consume a study pudding that will be used to deliver a low and a high dose fiber product. Blood samples will be collected to measure background levels of metabolites. At day 0 participants will consume a low dose study product and day 6 the high dose study product and provide blood samples over an 8 hr period after study product consumption, to be followed by a 24 hr blood sample and 48 hr blood sample. Additionally following the low / high dose study product 24 and 48 h urine samples will be collected.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.50 - 29.99
* non Tobacco or vaping user
* non-user of hemp products within 12 months of first visit
* Willing to stop dietary supplement use within 7 days of visit
* Generally heathy

Exclusion Criteria:

* History or presence of clinically important disorders that may affect subjects ability to participate in the study
* Clinically important GI conditions that potentially interfere with evaluation of study product
* Uncontrolled hypertension or unstable use of antihypertensives
* Recent antibiotic use
* extreme dietary habits
* recent or currently on weight loss regimen
* Known allergy or sensitivity to the study products
* History or presence of cancer in prior 2 years, except for non-melanoma skin cancer
* History of any major trauma or major surgical event within 2 months of first visit
* Pregnancy or willing to become pregnant during study
* Alcohol abuses
* Exposure to any non-registered drug product within 30 days prior to first visit

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Blood concentration of phenolics from 0 to 8 hours | 0 to 8 hours after consumption

SECONDARY OUTCOMES:
Blood concentration of phenolics 0 to 24 hours | 0 to 24 hours after consumption
Urine concentration of phenolics 24 and 48 hours after consumption | cumulative total phenolics at 24 and 48 hours
Concentration of Phenolic metabolites in blood and urine | Blood concnetrations at 0 to 8 hours post consumption and cumulative urine concentration 24 hours and 48 hours post consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Biofortis, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No